CLINICAL TRIAL: NCT05178680
Title: Impact of the Combination of Music and Relaxing Light on the Patient's Anxiety Postoperatively After Cardiac Surgery in the Intensive Care Unit: Randomized Pilot Study.
Brief Title: Combination of Music and Relaxing Light on the Patient's Anxiety After Cardiac Surgery in the Intensive Care Unit
Acronym: RéaRelax
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RéaRelax
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Heart; Surgery, Heart, Functional Disturbance as Result; Anxiety; Pain, Postoperative; Delirium
Keywords: unit intensive care; heart surgery; anxiety; pain; delirium; non medicinal technique; music; light
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative; Delirium; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- relaxation session combining music and soft light (Experimental)
  Interventions: Other: relaxation session combining music and soft light
- usual rest session (No Intervention)

INTERVENTIONS:
Other: relaxation session combining music and soft light — The caregiver will install a device consisting of a light bubble column, a multicolored light projector, and relaxing music chosen by the patient from a proposed panel. This session will last 30 minutes the day after the surgery
  Arms: relaxation session combining music and soft light

SUMMARY:
Cardiac surgery is not trivial. It requires opening the thorax in certain indications: coronary artery bypass grafting, valve replacements or plasties, aortic dissection, etc. These different procedures, both pre- and post-op, generate anxiety in the patient, the effects of which can be harmful to the recovery process and general well-being. It can be increased by the resuscitation environment during the immediate postoperative management. This environment also favors the development of delirium. It is possible to improve this environment by using non-drug and inexpensive techniques. Indeed, making the stay in the ICU better while respecting the safety of the patient and the efficiency of the care, could reduce anxiety as well as the appearance of delirium. Studies have been carried out on the effectiveness of music in health care with a positive impact on anxiety and pain.

The proposed study aims to evaluate the implementation of relaxation moments adapted to the resuscitation sector from the day after surgery. They target the senses available and accessible at that moment, such as hearing (relaxing music chosen by the patient will be played) and sight (a multi-effect light projector and a bubble column will be deployed). Environmental stressors will be minimized, while maintaining an optimal level of safety.

The primary objective is to compare anxiety before and after the first session in cardiac surgery patients in the cardiothoracic and vascular surgery (CCTV) resuscitation unit between the group with the usual rest session and the group with the rest session combining soft music and light.

The secondary objectives are based on an evaluation of anxiety over different time periods, patient comfort, occurrence of postoperative delirium, patient pain, average length of stay (LOS).

This is a pilot, comparative, monocentric, randomized, interventional research with minimal risks and constraints in 2 parallel groups. 110 patients will be included over a period of 12 months In the experimental group, once a day, a relaxation session with the association of soft music and light will be proposed by adapting the environment of the patient's resuscitation room. The control group will have the usual rest session.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient going for scheduled or semi-emergency cardiac surgery: any patient who had an anesthesia consultation for cardiac surgery ≥ 48 hours before surgery (according to the recommendations of the French Society of Anesthesia and Intensive Care)
* Patient affiliated or beneficiary of a social security plan;
* Patient without guardianship or curatorship, or subordination.
* Informed consent signed by the patient after clear and fair information about the study

Exclusion Criteria:

* Deaf and/or blind patient
* Patients with a history of delirium or proven dementia.
* Persons benefiting from enhanced protection, i.e. minors, persons deprived of their liberty by a judicial or administrative decision, adults under legal protection (guardianship and trusteeship) and finally patients in a vital emergency situation.
* Pregnant or breastfeeding women, women of childbearing age who do not have effective contraception (hormonal/mechanical: per os, injectable, transcutaneous, implantable, intrauterine device, or surgical: tubal ligation, hysterectomy, total ovariectomy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-05-13 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
State Tait Anxiety Inventory Measure before and after the 1st session in patients undergoing cardiac surgery, in the intensive care unit for cardio thoracic and vascular surgery | 5 days
  the difference in the result of the anxiety assessment before and after the 1st session with state-Trait Anxiety Inventory Y

CONTACTS AND LOCATIONS:
Overall Officials: GIRAULT Aurélie, Principal Investigator — CHU Poitiers
Locations (1):
- Réanimation cardio-thoracique, Poitiers, France